CLINICAL TRIAL: NCT02497885
Title: Seroprevalence of IgG Antibodies to Middle East Respiratory Syndrome Coronavirus in Asymptomatic Healthcare Workers After Treatment of Confirmed MERS Patient
Brief Title: Seroprevalence of MERS-CoV IgG in Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Hee Jung Choi, Professor, Ewha Womans University Mokdong Hospital
Other Study IDs: KMSG_HCW_IgG
Record Dates: First submitted 2015-07-06; First posted 2015-07-15 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Coronavirus Infections
Keywords: MERS; healthcare personnel
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthcare personnel group: healthcare worker who was exposed to confirmed MERS patients, irrespective of adequate personal protective equipment.

SUMMARY:
The investigators aim to do serosurvey of healthcare-personnel who had participated in treatment of confirmed patients of Middle-East respiratory syndrome. The investigators collected the base-line (pre-exposure) serum of healthcare-personnel in a few centers, and will collect the post-exposure serum from about 25-30 centers in which confirmed MERS patients had been treated.

The investigators will deduct the seroprevalence of MERS-CoV IgG among the healthy healthcare-personnel, and calculate the sero-conversion rate if possible. The investigators will subdivided the seroprevalence according to the degree of exposure and preparedness of personal protective equipment.

DETAILED DESCRIPTION:
We aim to deduct the seroprevalence of healthcare-personnel (HCP) who had participated in treatment of confirmed patients of Middle-East respiratory syndrome.

In first step, we collected the base-line (pre-exposure) serum from the HCP who worked in the hospitals in which confirmed MERS patients were treated. Pre-exposure serum was collected in a few centers. If the serum was drawn within 3 weeks from initial exposure, then the serum was considered adequate as pre-exposure. (Because, antibody against the MERS-CoV would be produced after more the 17-21 days of exposure). The serum was frozen.

In second step, we will collect the post-exposure serum from the HCP who worked in the hospitals in which confirmed MERS patients were treated or detected. We plan to include 25-30 centers. The timing of sample collection is 6-8 weeks after last contact with confirmed MERS patients. The serum will also freeze.

In third step, we will assay the presence of antibody in collected sample. We will use MERS-CoV ELISA kit (EUROIMMUNE co.) as screening test and MERS-CoV IFA kit (EUROIMMUNE co.) as confirm test.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare-personnel who are working for hospitals in which confirmed MERS patients were treated or detected
* Close contact with confirmed patient(s).
* Agree to informed consent

Exclusion Criteria:

* disagree to consent
* confirmed MERS patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthcare-personnel
Sampling Method: Non-Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
IgG(+) | up to 4-5 month
  MERS-CoV IgG(+)

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jung Choi, MD, PhD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha womans university mokdong hospital, Seoul, South Korea